CLINICAL TRIAL: NCT03659331
Title: A Controlled Study of Potential Therapeutic Effect of Oral Zinc in Manifesting Carriers of Wilson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Elon Pras (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Elon Pras, head of The Institute of Human Genetics, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4987-18-SMC
Record Dates: First submitted 2018-08-28; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Zinc; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: A model based on the assumption that at least 50 subjects will be recruited, and assuming that 50% of the patients will have a significant reduction of liver enzymes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- unexplained elevation of liver enzymes (Experimental): patients over the age of 18 referred for unexplained elevation of liver enzymes and carry a single mutation in the ATP7B gene. After a washout period of 3 months these patients will be re-checked for liver enzymes and if high will receive zinc therapy at a dose of 300 mg / day for 6 months, after which the liver enzymes will be checked again.
  Interventions: Dietary Supplement: Zinc

INTERVENTIONS:
Dietary Supplement: Zinc — blood tests will be performed: GGT SGOT, SGPT, LDH, A.P. Direct and indirect bilirubin, blood proteins, cholesterol, P.T. and a complete blood count.
  Other Names: blood tests

SUMMARY:
The assumption is that in some of the carriers, the increase in enzymes reflects tissue damage due to excess copper. The reduction of the amount of copper absorbed will decrease excess copper in the liver, which will result in a decrease in the level of liver enzymes. Zinc causes the induction of metalothionines in the intestine, which in turn prevents absorption of copper from the digestive system. Zinc administration in Wilson's patients causes the depletion of copper deposits and constitutes one of the cornerstones in the treatment of this disease.

DETAILED DESCRIPTION:
The research group is composed of patients over the age of 18 referred for unexplained elevation of liver enzymes and carry a single mutation in the ATP7B gene. After a washout period of 3 months these patients will be re-checked for liver enzymes and if high will receive zinc therapy at a dose of 300 mg / day for 6 months, after which the liver enzymes will be checked again.

ELIGIBILITY:
Inclusion Criteria:

patients over the age of 18 unexplained elevation of liver enzymes patients that carry a single mutation in the ATP7B gene.

-

Exclusion Criteria:

na

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
measurement of liver enzymes in blood tests | 9 months
  A model based on the assumption that at least 50 subjects will be recruited, and assuming that 50% of the patients will have a significant reduction of liver enzymes, is statistically significant and supports the association between a single mutation in the ATP7B gene and liver injury.

CONTACTS AND LOCATIONS:
Overall Officials: Elon Pras, Prof, Principal Investigator — The Institute of Human Genetics, Sheba Medical Center, Israel